CLINICAL TRIAL: NCT01984944
Title: Characterisation of Circadian Rhythm in Autistic Spectrum Disorder : a Clinical, Biochemical and Genetic Study
Brief Title: Characterisation of Circadian Rhythm in Autistic Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Henri Mondor University Hospital (Other); Albert Chenevier Hospital (Department of Psychiatry) (Unknown); Hopital Universitaire Robert-Debre (Other); Pasteur Institute (Cognitive Function and Human Genetic) (Unknown); Fondation FondaMental (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P081103; 2009-011842-24 (EudraCT Number)
Record Dates: First submitted 2013-10-29; First posted 2013-11-15 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Autistic Disorder
Keywords: circadian rhythm
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autistic Patient (Other): * 50 adults
  * 25 childs
  Interventions: Other: Autistic functional exploration
- Controls (Other): * 50 adults
  * 25 childs
  Interventions: Other: Control functional exploration

INTERVENTIONS:
Other: Autistic functional exploration — * 50 adults with urinary sample, core body temperature rhythm, Circadian rhythms assessed with actometer
  * 25 childs with urinary sample, Circadian rhythms assessed with actometer
  Arms: Autistic Patient
Other: Control functional exploration — * 50 adults with urinary sample, core body temperature rhythm, Circadian rhythms assessed with actometer
  * 25 childs with urinary sample, Circadian rhythms assessed with actometer
  Arms: Controls

SUMMARY:
Autism spectrum disorders (ASDs) are complex neurodevelopmental conditions characterized by deficits in social communication, delay in language and repetitive behaviors. Results from genetic studies reveal one pathway associated with susceptibility to ASDs, which includes synaptic cell adhesion molecules. Among the factors that could modulate this pathway are the genes controlling circadian rhythms. Sleep disorders and low melatonin levels are frequently observed in ASDs. Thus investigator will characterize the circadian rhythms of patients with ASD and search for circadian rhythms genes polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with autistic spectrum disorders
* At least 6 years old
* Membership of a social security scheme
* Informed consent signed by the patient or both holders of parental authority if the subject is a minor, or by a guardian if the subject is under guardianship

Exclusion Criteria:

* Recent sleep symptoms
* Incapacity to keep rested for 24 hours

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Urinary sulfatoxymelatonin secretion | The determination will be performed at 14 days ( child)
Urinary sulfatoxymelatonin secretion | The determination will be performed at 21 days ( adults)

SECONDARY OUTCOMES:
Core body temperature rhythm | The determination will be performed at 5 days (adult)
Circadian rhythms assessed with actometer | The determination will be performed at 14 ( child) and 21 days (adult)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DROUOT, MCU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France